CLINICAL TRIAL: NCT05206669
Title: TESTING MESSAGES TO PROMOTE USE OF AN HPV ONLINE INTERVENTION
Brief Title: Testing Messages to Promote HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 16-0447
Record Dates: First submitted 2021-12-17; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Behavior, Information Seeking; Intention; Vaccine Hesitancy
Keywords: HPV vaccine; Vaccine intention
MeSH Terms: conditions — Information Seeking Behavior; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: The current study employed a 2 x 3 mixed factorial design. Participants consisted of two groups: 1) Hispanic or Latino parents of adolescents (age 11-17), and 2) Hispanic or Latino young adults (age 18-26). Participants were randomly assigned to one of three message conditions: cancer, genital warts, or control messages.
Who Masked: Participant
Masking Description: Participants were not informed of the study design and were unaware of the other message conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cancer Messages - Young Adults (Experimental): Messages providing information about the use of HPV vaccines to prevent cancer.
  Interventions: Behavioral: Health Messages
- Cancer Messages - Parents of Adolescents (Experimental): Messages providing information about the use of HPV vaccines for their adolescent children to prevent cancer.
  Interventions: Behavioral: Health Messages
- Genital Wart Messages - Young Adults (Experimental): Messages providing information about the use of HPV vaccines to prevent genital warts.
  Interventions: Behavioral: Health Messages
- Genital Wart Messages - Parents of Adolescents (Experimental): Messages providing information about the use of HPV vaccines or their adolescent children to prevent genital warts.
  Interventions: Behavioral: Health Messages
- Control Messages - Young Adults (Active Comparator): Messages providing information about HPV vaccines that did not mention prevention of other diseases or conditions.
  Interventions: Behavioral: Health Messages
- Control Messages - Parents of Adolescents (Active Comparator): Messages providing information about HPV vaccines for their adolescent children that did not mention prevention of other diseases or conditions.
  Interventions: Behavioral: Health Messages

INTERVENTIONS:
Behavioral: Health Messages — Brief messages providing information about the effectiveness of HPV vaccines. Messages included embedded links where participants could find more information.

SUMMARY:
Human papillomavirus (HPV) is the most common sexually transmitted infection worldwide. Hispanic women have the highest rates of HPV-related cervical cancer compared to all other groups in the U.S. Previous research has delineated several unique barriers to HPV vaccination among Hispanic women, suggesting that interventions that focus on addressing these barriers may improve HPV vaccination compliance in this population. To address some of these unique barriers, an online tailored messaging intervention was developed and tested. Initial analyses demonstrate that participants exposed to an online intervention demonstrated higher intentions to vaccinate for HPV after viewing the informational materials. The next phase of the project will be comprised of promoting use of the online intervention to the general public through the use of theory-based, pretested messages delivered via advertisements on Facebook and Twitter. Specifically, messages will be targeted based on differences between Hispanic parents of adolescents and Hispanic young adults. Previous research has explored the use of the Extended Parallel Processing Model as a theory to guide messages designed to promote health behaviors. The current study extends this work in the area of HPV prevention. Specifically, it seeks to examine the use of this theory as a means to stimulate information seeking behavior in the form of use of the previously developed online intervention that provides information about HPV. We also hope to make a significant contribution to research demonstrating the importance of targeting messages based on differences in population characteristics. Additionally, this study seeks to build on research examining the use of social media sites as a means for implementing health interventions and promoting positive health outcomes. Ultimately, the current study seeks to improve both the HPV vaccination decision-making process and HPV vaccination rates. If this was achieved among the Hispanic population it could substantially decrease disparities in cervical cancer and other HPV-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* For parents eligibility criteria were being: 1) of Hispanic or Latino origin, 2) 18 years or older, 3) a parent or guardian of a child ages 11-17 who had not been vaccinated for HPV.
* For young adults eligibility were being: 1) of Hispanic or Latino origin, 2) 18-26 years of age (vaccine eligibility at the time of data collection, and 3) having not been vaccinated for HPV.

Exclusion Criteria:

* Being under 18 years of age
* Not identifying as Hispanic or Latino
* For parents, having no children ages 11-17 or having only children already vaccinated for HPV
* For young adults, having already been vaccinated for HPV or no longer being eligible due to age (>26)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-03-05 (Actual); Study Completion 2017-03-05 (Actual)

PRIMARY OUTCOMES:
Intention to Seek Information - 1 | 1 day (one time while participants viewed the brief intervention.)
  Hyperlinks were embedded in intervention messages where participants were told they could find more information about HPV. A click on the link was considered intention to seek information. Not clicking on the link was considered no intention to seek information.
Intention to Seek Information - 2 | Outcome was measured one time immediately post-intervention via the post-survey items described to assess their degree of intention.
  Intention to Seek Information survey items measure participants likelihood to seek information about HPV. Survey items included a Yes-No response to the statement "I intend to look for more information about the HPV vaccination within the next 30 days." Those who answer "Yes" were then shown a series of questions prompting them to indicate their likelihood of seeking more information about the HPV vaccination from their "doctor or healthcare provider," "a friend of family member," "the Internet," and "other sources." Responses were measured on a 7-point Likert-type scale that ranged from Very Likely to Very Unlikely. Those who answered "No" were shown the question "Which of the following best represents your reason for not seeking information about the HPV vaccine?". Responses included 1) low interest in the topic, 2) already well informed on the topic, 3) topic is not relevant to me, and 4) information on this topic is upsetting to me.

SECONDARY OUTCOMES:
Intention to Vaccinate for HPV | Outcome was measured one time immediately post-intervention via the post-survey items described to assess their degree of intention
  Intention to Vaccinate for HPV measures participants willingness to vaccinate for HPV. It was measured using a single item stating "I intend to get vaccinated against HPV within the next 6 months." Reponses were measured on a 7-point scale ranging from "Strongly agree" to "Strongly disagree."

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reno JE, Dempsey AF. Promoting HPV vaccination among Latinx: an application of the extended parallel processing model. J Behav Med. 2023 Apr;46(1-2):324-334. doi: 10.1007/s10865-022-00293-7. Epub 2022 Feb 18. PMID 35178652